CLINICAL TRIAL: NCT02556541
Title: Ultrasound-guided Peripheral Vascular Access in Children - a Single- Blind, Randomized, Cross-over Trial
Brief Title: Ultrasound-guided Peripheral Vascular Access in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Model: Crossover | Purpose: Supportive Care
Other Study IDs: 1-10-72-94-15
Record Dates: First submitted 2015-09-15; First posted 2015-09-22 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2015-04

CONDITIONS: Ultrasonography; Vascular Access Devices; Pediatrics

INTERVENTIONS:
Procedure: IV puncture guided by ultrasound

SUMMARY:
The purpose of this investigation is to conduct a randomized, patient-blinded prospective controlled trial comparing peripheral intravenous cannulation in children done by:

1. Conventional landmark cannulation where the intravenous cannulation is done by direct visual guidance or palpation or a combination thereof.
2. Ultrasound guided cannulation by means of DNTP.

The investigators hypothesize that with ultrasound-guided peripheral intravenous cannulation the first-attempt success rate will be significantly higher than by the conventional landmark cannulation technique.

ELIGIBILITY:
Inclusion Criteria:

* Requirement for anaesthesia before MRI or operation.
* Routine need of peripheral intravenous cannulation.
* Age 0- 3 years at the date of MR scan

Exclusion Criteria:

* Lack of consent
* Emergency patients needing immediate operation or scan.

Max Age: 3 Years | Sex: All
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
First attempt success | Intraoperative
  Succes rate of first attempt cannulation for ultrasound and traditional method will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Intensive Care, Aarhus, Denmark